CLINICAL TRIAL: NCT06357156
Title: Evaluating the Topographic and Quantitative Differences of the Mandibular Symphysis Area Between Males and Females Egyptians Using CBCT Scans: a Cross-sectional Study
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Passant Yusuf Abulabas, assistant lecturer, Cairo University
Other Study IDs: ORAD-621
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Mandibular Symphysis, Block Bone Graft, Mandibular Incisive Canal, and CBCT

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- males age range 18-35
  Interventions: Radiation: CBCT
- males age range 36- 55
  Interventions: Radiation: CBCT
- males age range 56-75
  Interventions: Radiation: CBCT
- females age range 18-35
  Interventions: Radiation: CBCT
- females age range 36- 55
  Interventions: Radiation: CBCT
- females age range 56-75
  Interventions: Radiation: CBCT

INTERVENTIONS:
Radiation: CBCT — The data collection will be obtained from the data base available at the department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University. CBCT images will be obtained from Egyptian patients who were referred to the CBCT unit in oral and maxillofacial radiology department for different purposes.

SUMMARY:
Retrospective Data Analysis will be performed after the CBCT images are pooled from the computer database.

* Exposure parameters of the scans will vary depending on patients' sizes (according to the manufacturer's recommendations).
* Images showing lower anterior mandibular teeth with 0.2 -0.4 voxel sizes will be reviewed.
* The topography and the quantity of the mandibular symphysis area will be assessed through the different planes: sagittal, coronal and axial cuts as well as assessing the prevalence of MIC and its distance from inferior border of the mandible if detected. Correlation of results according to gender and age (3 age sub-groups per gender:18-35, 36- 55, 56-75).
* CBCT images will be interpreted by oral and maxillofacial radiologist; blinded from demographic data of the patients.
* radiologist (Principle investigator) will evaluate the images for assessing the topography and quantity of bone in symphysial area through measuring dimensions of mandibular symphysis. Then will re-evaluate twice with a time lag of two weeks between the two reading sessions. The assistant supervisor will evaluate percentage of the scans. Any disagreement will be solved by consensus between the two observers.
* The measurements will be carried out by the principle observer (PY) and will be repeated 2 weeks later for intra-observer reliability assessment.
* Mandibular scans will be collected from planmeca machine, with 0.2-0.4 voxel size to be viewed on Romexis software to do the measurements of mandibular symphysis. Vertical height will be measured from the apices of anterior teeth to inferior border of the mandible from the sagittal and coronal cuts with the orientation lines parallel to the buccal cortical plate. Also, the sagittal cuts will be used to determine the depth of the labial bone, from the apices of anterior teeth the labial cortical plate with the orientation lines parallel to the buccal cortical plate (Safi, Yaser et al.,2021) Whilst horizontal dimension (width) will be measured along the outer surface of the labial cortical bone, which is determined from the inter-foraminal distance. 3D slicer software will be used for this curved measurement on the axial plane, since Romexis software can only do the linear and angular measurements (Lee , Kim et al, 2014).

Also, the sagittal reformatted cuts will be used for the determination of the topography of bone in symphysial area; either class I, II or III (Jussara Constantino, et al., 2018) Radiographs showing the different topographic types Radiograph A: Type I, B: Type II and C: Type III

• Through scrolling in sagittal, coronal cuts and the reformatted panoramic view the prevalence of mandibular incisive nerve will be detected (Borghesi, Andrea et al., 2022).

After collecting the whole data, statistically will be correlated to the age and gender.

ELIGIBILITY:
Inclusion Criteria:

1. patients' age between (18-75) years, so that the anatomical features of the permanent dentition could be evaluated.
2. Mandibular CBCT images with fully or partially edentulous anterior teeth.
3. No history or presence of any pathological condition in the mandible

Exclusion Criteria:

1. Poor image quality
2. presence of artifact that impairs the diagnostic quality
3. Presence of any pathological condition in the mandible

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: A total sample of 222 mandibular CBCT scans belonging to Egyptian individuals will be included. The sample size will be sub-grouped to 3 age groups per each gender.
  The data collection will be obtained from the data base available at the department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University. CBCT images will be obtained from Egyptian patients who were referred to the CBCT unit in oral and maxillofacial radiology department for different purposes.
Sampling Method: Probability Sample
Enrollment: 222 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Effect of gender on the mean height of basal bone in the symphysial area | 1 year
  Oblique Reformatted cuts Built-in measuring tool (ruler) (Romexis software) in mm

SECONDARY OUTCOMES:
Effect of gender on quantity of the bone in symphysial area: *depth of the bone *width of the bone | 1 year
  Oblique Reformatted cuts Built-in measuring tool (ruler) (Romexis software) (3D-slicer software) in mm
Effect of gender on topography of the bone in symphysial area | 1 year
  Categorical assessment according to Locks, Bruna Jussara Constantino, et al., 2018 (class I,II or III)/Categorical nominal data (%)
Effect of age on quantity of the bone in the symphysial area | 1 year
  Oblique Reformatted cuts Built-in measuring tool (ruler) (Romexis software) (3D-slicer software) in mm
Effect of age on topography of the bone in symphysial area | 1 year
  Categorical assessment according to Locks, Bruna Jussara Constantino, et al., 2018 (class I,II or III)/Categorical nominal data (%)
Prevalence of mandibular incisive canal | 1 year
  Subjective judge of the radiologist using Oblique Reformatted cuts/present or absent

IPD SHARING:
Plan to Share IPD: Undecided